CLINICAL TRIAL: NCT04721535
Title: A Randomized Double-blinded Controlled Clinical Trial of DWJ1248 in Prevention of COVID-19 Infection After the Exposure of SARS-COV-2
Brief Title: A Study of DWJ1248 in Prevention of COVID-19 Infection After the Exposure of SARS-COV-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination of study due to sponsor's internal decision
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DW_DWJ1248303
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Covid19; SARS-COV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1248 (Experimental): Camostat mesilate 200mg
  Interventions: Drug: DWJ1248
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWJ1248 — Orally, 1 tablet of DWJ1248 TID, up to 14 days
  Arms: DWJ1248
Drug: Placebo — Orally, 1 tablet of placebo TID, up to 14 days
  Arms: Placebo

SUMMARY:
To evaluate the prevention of SARS-COV-2 infection after administration of DWJ1248 in person who contact from COVID-19 confirmed patient compared to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19 as of the signed date in written consent
* Subjects in self-quarantine who contact from COVID-19 confirmed patient
* Subjects who have COVID-19 negative RT-PCR result
* Subjects with no symptoms of COVID-19

Exclusion Criteria:

* Subjects who cannot orally administer the investigational products
* Subjects who need administration of immunosuppressants
* Subjects who are allergic or sensitive to investigational products or its ingredients
* Subjects who have a history of drug and/or alcohol abuse within 12 months before screening
* Subjects who have been identified with uncontrolled concomitant diseases or conditions, including significant mental illness and social conditions, that may affect compliance with clinical trial procedures according to the determination of the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with COVID-19 | Up to 14 days
  positive result in RT-PCR test

SECONDARY OUTCOMES:
Percentage of subjects with hospitalization | Days 3, 7, 14, and 28
  hospitalization due to COVID-19
Percentage of subjects who experience intensive care unit (ICU) | Days 3, 7, 14, and 28
  ICU requirement due to COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No